CLINICAL TRIAL: NCT01957410
Title: An Open-Label and Double-Blind Study to Investigate Evoked Potentials as Markers of Ketamine-induced Cortical Plasticity in Subjects With Major Depressive Disorder
Brief Title: A Study to Investigate Evoked Potentials as Markers of Ketamine-induced Cortical Plasticity in Patients With Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical Team decision to terminate the study after the results from Cohort 1 did not support conducting Cohort 2.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR102607; KETIVTRD2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Ketamine; Evoked potentials; Somatosensory evoked potentials; Motor evoked potentials; Cortical plasticity
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine Intravenous (IV) (Experimental): Patients will receive a single IV dose of ketamine given as a continuous infusion.
  Interventions: Drug: Ketamine
- Placebo Intravenous (IV) (Placebo Comparator): Patients will receive a single IV dose of placebo given as a continuous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — During Cohorts 1 and 2, a single ketamine 0.5 mg/kg dose will be given as a continuous IV infusion over 40 minutes by use of an electronic syringe infusion pump. The predefined dose and infusion rate/duration should not be adjusted. If a patient is unable to tolerate the study medication, the infusion should be stopped. Within 1 week of completion of the open-label treatment phase, participants can receive a single dose of ketamine 0.5 mg/kg administered as an IV infusion over 40 minutes during an optional open-label treatment phase.
  Arms: Ketamine Intravenous (IV)
Drug: Placebo — During Cohort 2, a single placebo dose will be given as a continuous IV infusion over 40 minutes by use of an electronic syringe infusion pump. Within 1 week of completion of the double-blind treatment phase, participants can receive a single dose of ketamine 0.5 mg/kg administered as an IV infusion over 40 minutes during an optional open-label treatment phase.
  Arms: Placebo Intravenous (IV)

SUMMARY:
To evaluate if somatosensory evoked potentials (SEPs) and motor evoked potentials (MEPs) obtained with electroencephalography (EEG) and electromyography (EMG) can be used to detect changes in cortical plasticity in responders to a single IV infusion of ketamine as compared to non-responders.

DETAILED DESCRIPTION:
This study will be conducted in patients with Major Depressive Disorder (MDD) and divided into 2 sequential cohorts. Cohort 1 will be conducted in 12 patients at a single center. For each patient, there will be up to 4 sequential phases: a screening phase of up to 6 weeks, an open-label treatment phase of up to 4 weeks, an optional open-label treatment phase of up to 1 week, and a follow-up phase of up to 1 week (if applicable). Cohort 2 will be conducted in 20 patients and will be a multicenter, double-blind (neither physician nor patient knows the treatment that the patient receives), randomized (the study drug is assigned by chance), placebo-controlled (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) design. For each patient, there will be up to 4 sequential phases: a screening phase of up to 6 weeks, a double-blind treatment phase of up to 4 weeks, an optional open-label treatment phase of up to 1 week, and a follow-up phase of up to 1 week (if applicable). The total study duration for each patient will be maximally about 12 weeks. Participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be medically stable
* Patient must meet Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV) diagnostic criteria for Major Depressive Disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the Mini International Psychiatric Interview (MINI)
* Patient must have had an inadequate response to at least 2 antidepressants, one of which is in the current episode of depression
* Patient must have an Inventory of Depressive Symptomatology 30-item Clinician-rated (IDS-C30) total score ≥ 34 at Screening and Day -1
* Women must be postmenopausal, surgically sterile, or, if heterosexually active, practicing a highly effective method of birth control
* Men who are heterosexually active with a woman of childbearing potential must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Patient has current signs and/or symptoms of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbances
* Patient has a primary DSM-IV diagnosis of current (active) generalized anxiety disorder (GAD), panic disorder, obsessive compulsive disorder (OCD), posttraumatic stress disorder (PTSD), anorexia nervosa, or bulimia nervosa
* Patient has a current diagnosis of bipolar disorder, mental retardation, or cluster b personality disorder (e.g., borderline personality disorders, antisocial personality disorder, etc)
* Patient has a current or prior diagnosis of a psychotic disorder or MDD with psychosis
* Patient has not responded to treatment with electroconvulsive therapy (ECT) in the current episode of depression
* Patient has suicidal ideation with intent to act, or has homicidal ideation/intent, during Screening phase per Investigator's clinical judgment
* Patient has any significant primary sleep disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants were enrolled, treated and completed the study.
Groups:
- Ketamine IV 0.5mg/kg: Participants received a single ketamine 0.5 milligram per kilogram (mg/kg) dose as a continuous Intravenous (IV) infusion over 40 minutes by use of an electronic syringe infusion pump on Day 1. Participants who responded continued the open-label treatment phase through Day 28 or until relapse, whichever occurred first. An additional single IV dose of ketamine 0.5 mg/kg was available during an optional open label treatment phase.
Period: Open Label
Arm/Group | Ketamine IV 0.5mg/kg
Started | 13
Completed | 13
Not Completed | 0
Period: Optional Open Label
Arm/Group | Ketamine IV 0.5mg/kg
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were received at least one dose of study drug.
Arm/Group | Ketamine IV 0.5mg/kg
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (11.45)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Region of Enrollment [Number; unit: participants]
  USA | 13

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Ketamine Responders and Ketamine Non-responders in the Change From Baseline in Somatosensory Evoked Potential (SEPs) Amplitudes at 4 Hours Postdose on Day 1
Description: SEPs are the electrical signals generated by the nervous system in response to somatosensory stimuli - typically through electrical stimulation of the median nerve. SEPs are read on the skull with electroencephalography (EEG). SEPs was recorded using a 64-channel EEG system at baseline (predose) and regularly after study drug administration. The change from baseline was calculated as post-baseline value minus baseline value for each participant. Since the number of participants at baseline differ from the number of participants at post-baseline measure (that is [i.e.] not all baseline values are paired), the mean change is not equal to the difference between the means at the two time points.
Time Frame: Baseline and Day 1 (4 hours postdose)
Population: Efficacy analysis set included all participants who received a dose of ketamine and who had at least 1 postbaseline value of SEP (P40).
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Ketamine IV 0.5mg/kg
Number analyzed (Participants) | 13
millivolts (mV)
  Responders: Baseline (n=9) | 1.83 (1.13)
  Responders: Day 1, 4 Hours (n=6) | 2.58 (1.24)
  Responders: Change from Baseline (n=6) | 0.47 (1.68)
  Non-Responders: Baseline (n=4) | 1.70 (1.10)
  Non-Responders: Day 1, 4 Hours (n=3) | 1.84 (1.48)
  Non-Responders: Change from Baseline (n=3) | 0.47 (0.43)

2. Primary Outcome: Comparison of Ketamine Responders and Ketamine Non-responders in the Change From Baseline in Motor Evoked Potential (MEPs) Amplitudes at 4 Hours Postdose on Day 1
Description: MEPs are generated when stimulation of the brain on the motor cortex (with Transcranial Magnetic Stimulation [TMS]) causes the spinal cord and peripheral muscles to produce neuroelectrical signals. MEPs are typically measured in the hand muscles. The Motor Evoked Response to Transcranial Magnetic Stimulation (TMS MEPs) was evaluated at baseline and regularly after study drug administration. Intracortical inhibition and facilitation was also evaluated using TMS. A figure-of-eight coil with external loop diameters of 9 cm was used to elicit motor responses in the contralateral first dorsal interosseus.
Time Frame: Baseline and Day 1 (4 hours postdose)
Population: Efficacy analysis set included all participants who received a dose of ketamine and who had at least 1 postbaseline value of MEP.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Ketamine IV 0.5mg/kg
Number analyzed (Participants) | 13
mV
  Responders: Baseline (n=9) | 0.874 (0.710)
  Responders: Day 1, 4 hour (H) (n=9) | 1.052 (0.867)
  Responders: Change from Baseline (n=9) | 0.179 (0.765)
  Non-Responders: Baseline (n=4) | 1.257 (1.055)
  Non-Responders: Day 1, 4H (n=4) | 1.197 (1.067)
  Non-Responders: Change from Baseline (n=4) | -0.060 (0.088)

ADVERSE EVENTS:
Time Frame: Up to 1 week after the last dose administration (6 weeks)
Arm/Group | Ketamine IV 0.5mg/kg
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine IV 0.5mg/kg (N=13)
Nausea (Gastrointestinal disorders) | 1 (1)
Infusion site bruising (General disorders) | 2 (2)
Bacterial vaginosis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Panic attack (Psychiatric disorders) | 2 (3)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was planned as open label treatment phase (Cohort 1) and double blind treatment phase (Cohort 2). However, study was terminated after completion of Cohort 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.